CLINICAL TRIAL: NCT00902876
Title: A Randomized Controlled Clinical Trial to Evaluate Safety and Effectiveness of CAF + Mucograft® Compared to CAF Alone in Patients With Gingival Recessions.
Acronym: MCT-Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10812-009
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2012-02

CONDITIONS: Gingival Recession
Keywords: root coverage; gingival recession; keratinized gingiva
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mucograft + CAF (Experimental): Mucograft in combination with coronally advanced flap (CAF)
  Interventions: Device: Mucograft
- CAF (Experimental): Coronally advanced flap (CAF) alone
  Interventions: Procedure: Coronally advanced flap (CAF)

INTERVENTIONS:
Device: Mucograft — Collagen Matrix for soft tissue regeneration
  Arms: Mucograft + CAF
Procedure: Coronally advanced flap (CAF)
  Arms: CAF

SUMMARY:
The purpose of this multi-center study is to determine the efficacy and safety of Mucograft® in combination with the coronally advanced flap (CAF) for the treatment of gingival recessions. It is assumed that the CAF combined with Mucograft® will result in improved outcome in terms percentage of root coverage and soft tissue thickness in comparison to CAF alone (control).

DETAILED DESCRIPTION:
Primary goals of mucogingival surgery have changed with time from maintaining gingival health and prevent further progression of the recession to providing predictable root coverage solving patients' esthetic demands.

Many surgical techniques have been utilized to restore gingival tissue dimensions including the use of autologous soft tissue graft. Longitudinal studies have shown that procedures using pedicle and free grafts are both effective for this purpose. However, since this technique uses epithelialized grafts, it generally results in compromised aesthetics ("patch-like area"). Alternatively free connective tissue grafts (CTG) are used providing similar predictability but resulting in better colour matching. Unfortunately, both techniques are associated with significant patient morbidity due to the wound at the palatal donor site. To avoid patient morbidity, acellular dermal allografts have been used as substitutes for palatal donor tissue, demonstrating the possible and promising use of allograft material. However, since the allograft material is derived from human cadavers; it is associated with ethical concerns and the risk of disease transmission.

In patients with a residual amount of keratinized tissue, the coronally advanced flap (CAF) - first introduce by Norber et al. (1926) - has been demonstrated to be very effective in treatment of multiple and single recessions with advantages in terms of aesthetics and morbidity. Although CAF is a safe and predictable approach for root coverage, the application of this surgical technique in conjunction with autologous or synthetic material was reported to enhance the probability to achieve complete root coverage in Miller Class I and II gingival recessions. A promising option to avoid patient morbidity and the use of autologous transplants or allografts is the use of collagen matrices from porcine origin, such as Mucograft®. Similar devices have been extensively used for guided tissue regeneration procedures. Mucograft® provides an ideal matrix for blood vessel and soft tissue ingrowth, which is likely to improve the results and the predictability of recession coverage procedure using the CAF.

ELIGIBILITY:
Inclusion Criteria:

* The patient (male or female) must be 18 years or older
* The patient must be a candidate for bilateral root coverage procedure
* Recession defects are Miller Class I-II and do not vary more than 2 mm.
* At least one mm keratinized tissue is present.
* Patient shows sufficient plaque control (FMPS < 20%).
* If patient is of child-bearing potential, the patient confirms not to be pregnant and agrees to take contraception for at least 6 months after surgery.
* The patient is able to comply with the study-related procedures such as exercising good oral hygiene and attending all follow-up procedures
* The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent.

Exclusion Criteria:

* Patient is a heavy smoker (> 10 cigarettes per day)
* Patient is an insulin dependent diabetic
* General contraindications for dental and/or surgical treatment are present.
* The patient has a history of malignancy, radiotherapy, or chemotherapy for malignancy within the past five years.
* The patient is pregnant or nursing
* The patient is taking medications or having treatments which have an effect on mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs).
* The patient has a disease, which affects connective tissue metabolism (e.g. collagenases).
* The patient is allergic to collagen.
* Patients have participated in a clinical trial within the last six months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
percentage of root coverage | 6 month

SECONDARY OUTCOMES:
gingival thickness | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Prof., Principal Investigator — Department of Periodontology, University Complutense Madrid, Spain; Soren Jepsen, Prof., Principal Investigator — Department of Periodontology, University of Bonn, Germany; Jan Wennström, Prof., Principal Investigator — Department of Periodontology, University of Gothenburg, Sweden; Giovanni Zucchelli, Prof., Principal Investigator — Department of Periodontology, University of Bologna, Italy; Lorenz Uebersax, Dr., Study Director — Geistlich Pharma AG, Wolhusen, Switzerland; Bernd Heinz, Dr, Principal Investigator — Private practice Hamburg, Germany; Massimo DeSanctis, Prof., Principal Investigator — Private Practice Firenze
Locations (1):
- Prof. Mariano Sanz, Madrid, Spain

REFERENCES:
- [Derived] Jepsen K, Stefanini M, Sanz M, Zucchelli G, Jepsen S. Long-Term Stability of Root Coverage by Coronally Advanced Flap Procedures. J Periodontol. 2017 Jul;88(7):626-633. doi: 10.1902/jop.2017.160767. Epub 2017 Mar 17. PMID 28304210